CLINICAL TRIAL: NCT00588406
Title: Emergency Department (ED) Use of Nebulized Budesonide as an Adjunct to Standardized Therapy in Acutely Ill Adults With Refractory Asthma: a Randomized, Double-blinded, Placebo-controlled Trial
Brief Title: Study of Budesonide as an Addition to Standard Therapy in Adult Asthmatics in the Emergency Room.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: AstraZeneca (Industry); Jacobi Medical Center (Other); Nassau University Medical Center (Other)
Responsible Party: Principal Investigator, Robert A Silverman, Physician, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 07.02.019
Record Dates: First submitted 2007-12-21; First posted 2008-01-08 (Estimated); Results first posted 2016-01-21 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2015-12

CONDITIONS: Asthma
Keywords: acute, emergency department
MeSH Terms: conditions — Asthma; Emergencies | interventions — Budesonide; Albuterol; Procaterol; Ipratropium; Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- B (Experimental): Budesonide, 2mg, 4 doses, plus standard care
  Interventions: Drug: Budesonide; Drug: albuterol; Drug: Ipratropium bromide; Drug: Prednisone
- P (Placebo Comparator): Placebo plus standard care
  Interventions: Drug: albuterol; Drug: Ipratropium bromide; Drug: Prednisone

INTERVENTIONS:
Drug: Budesonide — 2mg/dose by nebulizer, four doses over 3 hours
  Other Names: Pulmicort Respules
  Arms: B
Drug: albuterol — 2.5mg/dose by nebulizer, 7 doses over 6 hours
  Other Names: proventil; proair; ventolin; salbutamol
Drug: Ipratropium bromide — 2.5 mg, one dose
  Other Names: Atrovent
Drug: Prednisone — 60mg PO
  Other Names: deltasone

SUMMARY:
To determine whether adding nebulized inhaled steroids to the standard care of acutely ill ED patients with refractory acute asthma helps improve forced expiratory volume at one second (FEV1) and decrease the need for hospitalization.

DETAILED DESCRIPTION:
This is a randomized clinical trial studying the effect of nebulized budesonide (Pulmicort) in acutely ill adults presenting to the Emergency Department with severe asthma. Budesonide is an inhaled steroid FDA approved for the treatment of pediatric chronic asthma. ED entry criteria include hyporesponsiveness to nebulized beta-agonists and an FEV1<50% predicted. The trial will evaluate the efficacy of multiple doses of nebulized budesonide as an adjunct to a highly regimented standardized treatment protocol; standard care consists of bronchodilators (beta-agonists/anticholinergics), systemic steroids, and intravenous magnesium sulfate (if the FEV1<25% predicted). The primary efficacy endpoint will be the FEV1 4 hours after administration of the study intervention. An additional safety and efficacy endpoint will take place at 5 hours after study intervention. The treatments will be coupled with a protocol-defined assessment regimen, with endpoints measured before each treatment and on ED disposition (at 5 hours after study intervention).

ELIGIBILITY:
Inclusion Criteria:

* FEV1<50% predicted after bronchodilator therapy, age 18-60, presenting to an emergency department with acute asthma

Exclusion Criteria:

* other chronic lung disease, >15 pack years smoking

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2007-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Silverman, MD, Principal Investigator — Northwell Health
Locations (3):
- United States (3):
  - Nassau University Medical Center, East Meadow, New York
  - Long Island Jewish Medical Center, Queens, New York
  - Jacobi Medical Center, The Bronx, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- Budesonide: Budesonide, 2mg, 4 doses, plus standard care
  Budesonide: 2mg/dose by nebulizer, four doses over 3 hours
  albuterol: 2.5mg/dose by nebulizer, 7 doses over 6 hours
  Ipratropium bromide: 2.5 mg, one dose
  Prednisone: 60mg PO
- Placob: Placebo plus standard care
  albuterol: 2.5mg/dose by nebulizer, 7 doses over 6 hours
  Ipratropium bromide: 2.5 mg, one dose
  Prednisone: 60mg PO
Period: Overall Study
Arm/Group | Budesonide | Placob
Started | 46 | 49
Completed | 46 | 49
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo plus standard care
  albuterol: 2.5mg/dose by nebulizer, 7 doses over 6 hours
  Ipratropium bromide: 2.5 mg, one dose
  Prednisone: 60mg PO
- Total: Total of all reporting groups
Arm/Group | Budesonide | Placebo | Total
Number analyzed (Participants) | 46 | 49 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.2 (11.4) | 42.6 (11.4) | 40 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 22 | 51
  Male | 17 | 27 | 44
Race/Ethnicity, Customized [Number; unit: participants]
  White | 2 | 3 | 5
  Black | 28 | 18 | 46
  Hispanic | 12 | 20 | 32
  Other | 2 | 6 | 8
  Unknown | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 46 | 49 | 95
Forced expiratory volume at one second (FEV1) % predicted [Mean (Standard Deviation); unit: percent predicted of FEV1] | 29.5 (9.5) | 29 (8.1) | 29.2 (8.7)

OUTCOME MEASURES:

1. Primary Outcome: FEV1 Percent Predicted
Time Frame: 4 hours post-randomization
Measure: Mean (Standard Deviation); unit: percent predicted of FEV1
Arm/Group | Budesonide | Placebo
Number analyzed (Participants) | 46 | 49
percent predicted of FEV1 | 51.7 (16.8) | 52.6 (15.8)

2. Secondary Outcome: Hospitalization
Time Frame: 6 hours
Measure: Number; unit: percentage of participants
Arm/Group | Budesonide | Placebo
Number analyzed (Participants) | 46 | 49
percentage of participants | 39 | 39

ADVERSE EVENTS:
Arm/Group | Budesonide | Placebo
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/49
Other Adverse Events (participants affected / at risk) | 0/46 | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes